CLINICAL TRIAL: NCT03762798
Title: Can The Bridge Facilitate Successful Transition From Medication-Assisted Treatment (MAT) With Low-dose Sublingual Buprenorphine to Oral Naltrexone in Patients With Extended Remission of Opiate Use Disorder
Brief Title: Can The Bridge Transition Opiate Use Disorder Patients in Stable Recovery From Buprenorphine to Naltrexone
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Not able to enroll participants.
Sponsor: The Cleveland Clinic (Other)
Responsible Party: Principal Investigator, David Streem, MD, Principal Investigator, The Cleveland Clinic
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 18-863
Record Dates: First submitted 2018-11-28; First posted 2018-12-04 (Actual); Last update posted 2021-09-23 (Actual); Status verified 2021-09

CONDITIONS: Substance Use Disorders; Substance Abuse; Substance Use; Substance Dependence
Keywords: substance abuse; the bridge
MeSH Terms: conditions — Substance-Related Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Treatment (Experimental): All participants will receive the Bridge device.
  Interventions: Device: The Bridge

INTERVENTIONS:
Device: The Bridge — The Bridge (Also known as NSS-2) is a percutaneous, auricular field stimulator developed to alleviate pain through stimulation of peripheral cranial neurovascular bundles in the external ear that could potentially gain access to brain areas involved in fear, pain and nociception. After five days, the subject will return to the clinic for device removal and disposal.

SUMMARY:
This is an open-label, single center study of The Bridge in patients with sustained remission of opiate dependence on established, low-dose MAT with buprenorphine. A fixed number of patients will be admitted to the study.

DETAILED DESCRIPTION:
This is an open-label, single center study of The Bridge in patients with sustained remission of opiate dependence on established, low-dose MAT with buprenorphine. A fixed number of patients will be admitted to the study.

After determination that the subject meets the inclusion criteria and does not meet any of the exclusion criteria for the study, the subject will receive the device which will be applied in the clinical office setting on an outpatient basis. Buprenorphine MAT will be stopped immediately and the subject will be followed on an outpatient basis to ensure the process has been successful. The subject will have the option to return to the office for a follow-up assessment in 1-4 days after device application. Seven to ten days after the last dose of buprenorphine, a urine sample will be collected for drug testing and a prescription for naltrexone will be provided. Then three visits on a roughly monthly basis will be scheduled. At each visit a urine sample for drug testing will be collected. After three follow-up visits are completed, if the drug testing demonstrates continued sobriety, the subject will be released from the study and may or may not continue treatment with naltrexone.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of opiate use disorder, any severity
* Age range 18-99 years old
* Not pregnant or breastfeeding
* Able to understand and provide informed consent.
* Able to understand and speak the English language.
* At least one year of abstinence from drugs of abuse including, but not limited to, all opiates, cannabis, benzodiazepines, barbiturates, alcohol and cocaine.
* Use of nicotine is excluded from this criterion.
* Use of any prescribed, controlled substance, taken according to the prescribing instructions, for no more than seven consecutive days, at least three months prior to the subject's study enrollment, is excluded from this criterion.
* Taking dose of buprenorphine less than or equal to no more than 4 mg daily for at least three months prior to starting the study.
* In the case of Zubsolv rapid-dissolve tablets, equivalent daily dose maximum would be 2.9mg.
* In the case of Bunavail buccal film, equivalent daily dose maximum would be 2.1mg.
* At least one year of self-reported, established 12-step based recovery work, including
* Home group membership and regular attendance of two 12- step meetings per week
* Regular work with 12-step sponsor who can attest that the subject has worked through step nine of the twelve steps of Alcoholics Anonymous or a similar 12-step based mutual help organization.

Exclusion Criteria:

* Exhibits active psychosis or suicide ideation or is otherwise psychiatrically unstable.
* Positive Utox2 Immunoassay, Quantitative Pain Panel Liquid Chromatography/Mass Spectroscopy, or Ethylglucuronide test for any nonprescribed substance or medication.
* Meets criteria for any other active substance use disorder except nicotine
* Allergic to naltrexone or has any condition of such nature and/or severity that would clinically contraindicate the prescribing of naltrexone.
* Any condition that contraindicates the use of NSS-2 including hemophilia, cardiac pacemakers and psoriasis vulgaris.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2018-11-19 (Actual); Primary Completion 2020-10-25 (Actual); Study Completion 2020-12-01 (Actual)

PRIMARY OUTCOMES:
Primary Objective | Three Months
  Number of patients who complete three follow-up visits while taking naltrexone and produce entirely negative urine opiate screens during that period

CONTACTS AND LOCATIONS:
Overall Officials: David W Streem, MD, Principal Investigator — The Cleveland Clinic
Locations (1):
- Cleveland Clinic Lutheran Hospital, Cleveland, Ohio, United States

IPD SHARING:
Plan to Share IPD: No